CLINICAL TRIAL: NCT06709989
Title: Expositions Chimique et Microbiologique Des Femmes Dans Les Exploitations Bovines laitières
Brief Title: Chemical and Microbiological Exposure of Women on Dairy Cattle Farms
Acronym: DAISY-Expo
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Sponsor
Other Study IDs: C23-69; 2024-A00966-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2024-11-14; First posted 2024-11-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Occupational Exposure to Chemicals
Keywords: farmer; women; occupational exposure; chemicals; pesticides; biocides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, hair, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although professionals working on dairy cattle farms come into contact with a wide range of chemicals and microbiological agents, little is known about this possible exposure, which occurs a priori via inhalation and skin contact.

The aim of this research is to gain a better understanding of this chemical and microbiological exposure, and this research focuses in particular on professional women working on dairy cattle farms , who may be in charge of specific activities not commonly carried out by professional men.

Exposure to pesticides, antiparasitic products and disinfectants will be the first substances to be investigated, followed by other chemical or particulate compounds present in everyday and professional environments. Exposure to these compounds will be measured by their presence in the urine, feces (if possible) and hair of around 60 participating women, as well as in bovine tuft/head hair and, if possible, air samples taken in milking buildings.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman working on a dairy cattle farm in the "Grand Ouest" region of France
* Woman who speaks and understands French

Exclusion Criteria:

* working less than 20h/week in dairy farms
* Woman under legal protection
* unsigned consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women working on dairy cattle farms in West area of France
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Exposure to chemicals of women working on dairy farms | At inclusion and at the end of the follow-up (for hair-concentrations), and during specific periods of agricultural activities (with two 4-day periods of urine sample collection, one period of faeces collection, and one week of environmental sampling)
  Concentrations of pesticide molecules, biocides, disinfectants and microbiological agents, measured in
  * urines of professional women working on dairy farms,
  * the hair of professional women working on dairy farms,
  * faeces of professional women from dairy farms,
  * tuft/head hair from females in the herd on farms where female professionals work,
  * environmental samples of pesticide molecules (PPPs, pesticides), biocides, disinfectants and microbiological agents.

SECONDARY OUTCOMES:
Exposure to other chemicals | At inclusion and at the end of the follow-up (for hair-concentrations), and during specific periods of agricultural activities (with two 4-day periods of urine sample collection, one period of faeces collection, and one week of environmental sampling)
  Concentrations measured in urine, hair, feces, toupillon/head hair and environmental samples from the farm of other chemical compounds present in the participants' professional uses and environments.

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Chevrier, Principal Investigator — Inserm UMR1085 Irset
Locations (1):
- UMR1085 Irset, Rennes, France

IPD SHARING:
Plan to Share IPD: No
No or required a additional/new ethic authorization